CLINICAL TRIAL: NCT05261087
Title: Determining the Relationship Between Cognitive Function, Job Satisfaction and Sleep Quality in Factory Workers
Brief Title: The Relationship Between Cognitive Function, Job Satisfaction and Sleep Quality in Factory Workers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Nadiye Doğan, Physiotherapist, Izmir Bakircay University
Other Study IDs: 2021/346
Record Dates: First submitted 2022-01-26; First posted 2022-03-02 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Factory Workers
Keywords: Cognitive function , Sleep quality , Job satisfaction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Factory worker: Workers working in the TPI blade factory will be included in the study. Those working in the wind vane production at the factory are divided into departments. The 65.5 main mold workers, which will require the most attention, will be included in our work.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Individuals will not receive any interventions

SUMMARY:
The aim of this thesis study is to determine the relationships between cognitive functions, job satisfaction and sleep in individuals aged 30 and over.Individuals over the age of 30 working in the Sasalı branch of TPI Composite factory will be included in the study that we plan to do as a cross-sectional study.

Data will be collected at TPI Composite Factory Sasalı Branch Infirmary. Individuals' demographic information (age, height, weight) and cognitive functions, job satisfaction and sleep quality will be evaluated.

DETAILED DESCRIPTION:
By definition, cognition is collecting information from the environment; We can express this collected information as the ability to understand and interpret. cognitive functions; attention, short and long term memory, understanding, adaptation, language skills, decision making, abstract thinking, mathematical processing and executive functions.

executive functions; It is the ability of a person to plan purposeful action without any help, to interpret the information he has collected, and to always determine the next step in successive tasks.As the age progresses, the individual experiences problems in executive functions as a result of the change in the prefrontal region. Elderly individuals cannot concentrate and have problems solving problems. In addition, they show lower performance than young people in processing, using and strategizing. In other words, as the age progresses, it becomes more difficult to maintain attention in situations that require simultaneous processing and using several information.

This strain also affects the job satisfaction of individuals. The concept we call job satisfaction is a feeling that the employee experiences as a result of realizing that the work he does and the results of the work done coincide or allow them to overlap with his material and moral needs and personal value judgments.

The daily life activities of individuals whose job satisfaction is affected are also affected. In daily life activities, sleep is a physiological requirement for human beings. As a concept, sleep is a natural resting state in which the consciousness against external stimuli is completely or partially lost, the reaction power is weakened and all kinds of activities are greatly reduced.

Sleep needs differ according to age. Individuals experience sleep problems with advancing age. The depth of sleep decreases. The person wakes up at night and it becomes difficult to fall asleep again. The duration of night sleep decreases and the duration of sleep during the day increases.

When the literature is examined, there are many studies with young and middle-aged adults in studies on cognitive function.

Many studies have examined cognitive function and physical activity and sleep quality or physical activity and job satisfaction. No study evaluating the relationship between sleep quality and job satisfaction has been found in the literature.

In line with the studies in the literature, we thought that there would be a relationship between cognitive function, job satisfaction and sleep quality. Therefore, the aim of the study is to determine the relationships between cognitive functions, job satisfaction and sleep in individuals aged 30 and over.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Individuals aged 30 and over
* Being able to read and write Turkish

Exclusion Criteria:

* Conditions where cognitive functions are affected, such as dementia
* Being colorblind
* Having problems with speaking and understanding Turkish

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees in the 65.5 main mold divisions, who have been working in the factory over the age of 30 for more than 2 years, are included.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | At baseline
  We will evaluate the cognitive function with the CogniFit program.CogniFit General Cognitive Assessment (CAB) is the leading professional tool to help measure general cognitive well-being in children 7+ and adults using online cognitive tasks. The results of this neurocognitive test are useful for understanding the general cognitive state of the user and highlighting their strengths and weaknesses.This test battery has its own scoring system.
Sleep Quality | At baseline
  We will measure sleep quality with the Pittsburgh Sleep Quality Scale questionnaire.Subjective sleep quality of PUKI, sleep latency, sleep duration, habitual sleep efficiency, sleep disorder, use of sleeping pills, and daytime functioning It has 7 components. Some of the component specified with a single item, while some obtained by grouping the substance. Each The item is evaluated over 0-3 points and 7 The sum of the component score forms the total PUKI score. A high score indicates poor sleep quality.
Job satisfaction | At baseline
  We will measure job satisfaction with the Minnesota Job Satisfaction scale.The Minnesota Job Satisfaction Scale was developed by Dawis et al. in 1967 to determine the level of job satisfaction. The validity and reliability study in our country was carried out by Baycan and the scale was Cronbach's alpha value was found to be 0.77. internal and revealing external job satisfaction factors quintet consisting of 20 items with characteristics It is a Likert-type instrument. Neutral satisfaction score of the scale is 3. If the score from the scale is less than 3, the job job satisfaction is low, if it is greater than 3 is considered high.

CONTACTS AND LOCATIONS:
Overall Officials: Nadiye Doğan, Principal Investigator — Izmir Bakircay University
Locations (1):
- Izmir Bakircay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided